CLINICAL TRIAL: NCT02408276
Title: Longitudinal Evaluation of Hip Cartilage Degeneration: the Effect of Femoroacetabular Impingement
Brief Title: Longitudinal Evaluation of Hip Cartilage Degeneration: FAI
Status: Completed | Type: Observational
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2016-168; R01AR066069-01 (NIH)
Record Dates: First submitted 2015-03-27; First posted 2015-04-03 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-02

CONDITIONS: Femoroacetabular Impingement
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- dGEMERIC MRI technique: All tests and imaging are part of standard of care except follow up MRI, which will be performed in a random group from within the cohort and paid for through this grant.
  Interventions: Other: dGEMERIC MRI technique

INTERVENTIONS:
Other: dGEMERIC MRI technique — Patients will be treated surgically (hip arthroscopy) or nonoperatively (physical therapy) and pain medications as needed. For surgical patients, cartilage samples and surgeon operative reports will be a source of research. For both cohorts, MRIs, radiographs and patient reported outcome surveys will be additional research sources.
  All tests and imaging are part of standard of care except follow up MRI, which will be performed in a random group from within the cohort and paid for through this grant.

SUMMARY:
Femoroacetabular impingement (FAI) is one of the most common mechanisms leading to the development of early cartilage and labral damage in the non-dysplastic hip. Anatomic abnormalities of the proximal femur and/or acetabulum result in repetitive injury during dynamic hip motion, leading to abnormal regional loading of the femoral head-neck junction against the acetabular rim. The resulting damage to the cartilage, labrum, and surrounding capsular structures predispose the patient to developing hip pain and early osteoarthritic changes. Clinically, patients with FAI are a heterogeneous group, with a wide array of presentation from pain to instability that may or may not be related to activity. To date no studies have identified specific prognostic indicators associated with successful surgical treatment of FAI, leaving surgeons without adequate criteria to determine which patients are best suited for arthroscopy. The investigators propose to address this critical knowledge gap by identifying the patient characteristics and morphological features of the hip that are associated with the optimal clinical outcomes in patients undergoing hip arthroscopy or non-operative management for treatment of suspected FAI in order to establish a treatment algorithm for FAI patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients 35 years of age or younger enrolled in the HSS Hip Preservation Registry prior to September 30, 2016 with an MRI confirmed diagnosis of FAI will be eligible for inclusion in this study regardless of surgery status.
* Patients who agree to participate must complete a baseline questionnaire consisting of: 1) Modified Harris Hip Score (MHHS), an overall measure of hip condition; 2) the Hip Outcome Score (HOS), a measure developed specifically for younger active patients that measures quality of life and levels of sports and recreation; and 3) International Hip Outcome Tool (iHOT33), a newly developed hip specific outcome score, which measures a number of subscores relating to physical and social functioning with hip problems.

Exclusion Criteria:

* Patients over age 35 will be excluded as the focus of this study is early changes that may predispose to later degenerative changes.
* Patients undergoing revision hip arthroscopy as their first treatment in the Registry will not be eligible, as these are patients who have failed initial therapy.
* Patients with no complete questionnaires at any time point will be excluded.

Ages: 10 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 35 years of age or younger enrolled in the HSS Hip Preservation Registry prior to September 30, 2016 with an MRI confirmed diagnosis of FAI
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2014-12; Primary Completion 2025-12-18 (Actual); Study Completion 2025-12-18 (Actual)

PRIMARY OUTCOMES:
degree of cartilage degeneration | 5 years post operation
  degree of cartilage degeneration at 5 years post-presentation based on changes in cartilage morphology assessed using MRI (a two-dimensional fast spin echo sequence in the coronal and sagittal planes).

SECONDARY OUTCOMES:
dGEMERIC MRI measurements | 2 year post operation
  We will use MRI to localize and measure chondral and labral abnormalities to determine whether extent, location, or type of defect affect the outcome of hip arthroscopy in FAI.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Lyman, PhD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States